CLINICAL TRIAL: NCT07283003
Title: Prospective Randomized Study on the Necessity of Postoperative Stenting After Ureteroscopy (URS) for Ureteral Stones.
Brief Title: Evaluating Postoperative Pain After Ureterorenoscopy.
Acronym: STENTIMENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lukas J Hefermehl (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Sponsor-Investigator, Lukas J Hefermehl, Principal Investigator, Kantonsspital Baden
Organization: Kantonsspital Baden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00665
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Ureteral Stones
Keywords: pain app evaluation; ureterorenoscopy; double-J catheter; pain assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-Stent Group (Active Comparator): No postoperative double-J catheter following ureterorenoscopy.
  Interventions: Other: No Double-J catheter insertion
- Stent Group (Active Comparator): Routine postoperative double-J catheter insertion following ureterorenoscopy.
  Interventions: Procedure: Double-J catheter

INTERVENTIONS:
Other: No Double-J catheter insertion — Ureterorenoscopy without consecutive DJ-stent insertion.
  Arms: No-Stent Group
Procedure: Double-J catheter — Transurethral catheter insertion
  Arms: Stent Group

SUMMARY:
Comparison of routine postoperative stenting versus no stenting after ureterorenoscopy for ureteral stones to assess the necessity and impact on complication risk.

DETAILED DESCRIPTION:
After a ureteroscopy (URS) for the removal of ureteral stones, a double-J stent is routinely placed. Among other measures, this is intended to prevent pain caused by ureteral swelling, small residual fragments, blood clots, and potential drainage obstructions, which could lead to colic or fever. However, the evidence supporting the benefit of this practice is limited. At the same time, many patients report discomfort due to the stent (e.g., flank pain, dysuria, frequent urination, hematuria), which can significantly impact their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with ureteral stones scheduled for ureteroscopy (URS) and stone removal
* Previous pre-stenting
* Informed Consent as documented

Exclusion Criteria:

* Complex ureteral conditions (e.g., known ureteral strictures)
* Impacted stones
* Solitary kidney
* Patients with significant renal stones (>3mm)
* Previous ureteral surgeries (except endoscopic stone treatments)
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessment | up to 4 weeks postoperative
  Assessment of postoperative pain will be conducted using the Visual Analogue Scale (VAS) and the study-specific mobile application HEATMAP (Byldr GmbH, Switzerland). The primary outcome is the difference between the pain scores recorded by the VAS and those recorded by the HEATMAP application at predefined postoperative time points [both measured on a scale from 1-10, with higher scores indicating greater pain].

SECONDARY OUTCOMES:
Length of stay [days] | During the hospital stay, on average 2 days
  Time from surgery to discharge in days [d]
Pain Assessment | pre-/peri-/postoperative
  Assessment of pain level via Visual Analogue Scale (VAS), scale [1-10, higher scores indicates greater pain]
Pain Management | pre-/peri-/postoperative
  Documentation of pain management [according to the WHO Analgesic Ladder, 1-4, higher scores mean more intense pain treatment]
Secondary need of double-J catheter | up to 4 weeks postoperative
  (Please note, this applies only for patients that where in the intervention group.)
  Patient received a double-J catheter, binary [yes/no]
Procedure related readmissions | up to 4 weeks postoperative
  Readmission that can be linked to the URS, binary [Yes/No]
Procedure related reoperations | up to 4 weeks postoperative
  Reoperation that can be linked to the URS, binary [Yes/No]
Comprehensive Complication Index | up to 4 weeks postoperative
  Any complication that occurred within 30 days post surgery, Scale [from 0 (no complication) to 100 (death)]

CONTACTS AND LOCATIONS:
Overall Officials: Lukas John Hefermehl, PD Dr. med., Principal Investigator — Kantonsspital Baden AG
Locations (1):
- Kantonsspital Baden AG, Baden, Switzerland

IPD SHARING:
Plan to Share IPD: No
The data that will be recorded in this study will be available on reasonable request from the PI